CLINICAL TRIAL: NCT03873246
Title: Randomized, Controlled, Single-Masked Clinical Trial to Evaluate the Chronic Efficacy of OC-01 Nasal Spray on Signs of Dry Eye Disease (The MYSTIC Study)
Brief Title: Clinical Trial to Evaluate the Chronic Efficacy of OC-01 Nasal Spray on Signs of Dry Eye Disease (The MYSTIC Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-004
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OC-01 0.1%, 0.6 mg/ml (Active Comparator): OC-01 (varenicline) nasal spray, 0.6 mg/mL
  Interventions: Drug: OC-01 0.1% 0.6 mg/ml
- OC-01 0.2%, 1.2 mg/ml (Active Comparator): OC-01 (varenicline) nasal spray, 1.2 mg/mL
  Interventions: Drug: OC-01 (varenicline) nasal spray: 0.2 % (1.2 mg/ml)
- Placebo (Placebo Comparator): vehicle control
  Interventions: Other: placebo comparator

INTERVENTIONS:
Drug: OC-01 0.1% 0.6 mg/ml — OC-01 (varenicline) nasal spray: 0.1 % (0.6 mg/ml)
  Other Names: varenicline
  Arms: OC-01 0.1%, 0.6 mg/ml
Drug: OC-01 (varenicline) nasal spray: 0.2 % (1.2 mg/ml) — OC-01 (varenicline) nasal spray: 0.2 % (1.2 mg/ml)
  Other Names: varenicline
  Arms: OC-01 0.2%, 1.2 mg/ml
Other: placebo comparator — vehicle control
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the chronic safety and effectiveness of OC-01 Nasal Spray as compared to placebo on signs of dry eye disease (DED).

DETAILED DESCRIPTION:
Study OPP-004 was a Phase 2, single-center, randomized, masked (including subjects, Investigators, and study site personnel), placebo-controlled study designed to evaluate the safety and efficacy of OC-01 (varenicline) nasal spray in adult subjects with DED. The study planned to randomize approximately 120 subjects at least 22 years of age with a physicians' diagnosis of Dry Eye Disease and meeting all other study eligibility criteria to receive an application of OC-01 or placebo BID for 12 weeks. Subjects who terminated early during the application period were asked to complete safety assessments (if the subjects agree) prior to study exit. Subjects who were terminated early from the study were not replaced.

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to us an artificial tear substitute for dry eye symptoms within 6 months prior to Visit 1

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery (e.g. laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1
* Have a history or presence of an ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauswirth SG, Kabat AG, Hemphill M, Somaiya K, Hendrix LH, Gibson AA. Safety, adherence and discontinuation in varenicline solution nasal spray clinical trials for dry eye disease. J Comp Eff Res. 2023 Jun;12(6):e220215. doi: 10.57264/cer-2022-0215. Epub 2023 Apr 25. PMID 37096956
- [Derived] Quiroz-Mercado H, Hernandez-Quintela E, Chiu KH, Henry E, Nau JA. A phase II randomized trial to evaluate the long-term (12-week) efficacy and safety of OC-01 (varenicline solution) nasal spray for dry eye disease: The MYSTIC study. Ocul Surf. 2022 Apr;24:15-21. doi: 10.1016/j.jtos.2021.12.007. Epub 2021 Dec 15. PMID 34920097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%, 1.2 mg/ml | Placebo
Started | 41 | 41 | 41
Completed | 36 | 29 | 32
Not Completed | 5 | 12 | 9
Not completed — Adverse Event | 1 | 3 | 3
Not completed — Lost to Follow-up | 4 | 4 | 5
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Subjects in the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%, 1.2 mg/ml | Placebo | Total
Number analyzed (Participants) | 41 | 41 | 41 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (13.18) | 54.2 (11.77) | 55.8 (26.77) | 53.8 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 33 | 100
  Male | 9 | 6 | 8 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Other | 41 | 41 | 41 | 123
  Hispanic or Latino | 41 | 41 | 41 | 123
Baseline Schirmer's Test Score [Mean (Standard Deviation); unit: mm] — A Schirmer's test determines whether a person's eye produces enough tears to keep their eye moist and healthy. The amount of wetting is recorded by numbing the eye and placing a paper strip in the eye for 5 minutes. Schirmer's test scores range from 0-35 mm where a higher score is indicative of a better outcome.
  mm | 5.5 (2.46) | 5.4 (2.47) | 5.3 (2.04) | 5.4 (2.33)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Schirmer's Test Score From Baseline to 84 Days
Description: The Schirmer's test measures the amount of tears produced by numbing the eye and placing a paper strip in the eye for 5 minutes and distance of wetting was recorded following treatment with OC-01 or placebo. Schirmer's test scores range from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: Visit 1 (baseline) and Visit 6 (84 days)
Population: Subjects in the ITT Population-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Groups:
- OC-01 0.2%. 1.2 mg/ml: OC-01 (varenicline) nasal spray, 1.2 mg/mL
  OC-01 (varenicline) nasal spray: 0.2 % (1.2 mg/ml): OC-01 (varenicline) nasal spray: 0.2 % (1.2 mg/ml)
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%. 1.2 mg/ml | Placebo
Number analyzed (Participants) | 41 | 41 | 41
mm | 10.8 (1.29) | 11.0 (1.29) | 6.0 (1.29)

2. Other Pre Specified Outcome: Percent of Subjects Who Achieve ≥10 mm Improvement in Schirmer's Test Score From Baseline at Visit 6 (Day 84)
Description: as for outcome 1
Time Frame: Visit 1 (baseline) and Visit 6 (84 days)
Population: Subjects in the ITT-LOCF population
Measure: Count of Participants; unit: Participants
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%, 1.2 mg/ml | Placebo
Number analyzed (Participants) | 41 | 41 | 41
Participants | 15 | 20 | 10

3. Other Pre Specified Outcome: Percent of Subjects Who Achieve ≥10 mm Improvement in Schirmer's Test Score From Baseline at Visit 4 (Day 28)
Description: The Schirmer's test measures the amount of tears produced by placing a paper strip in the eye for 5 minutes and the distance of wetting was recorded following treatment with OC-01 or placebo. Schirmer's test scores range from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: Visit 1 (baseline) and Visit 4 (28 Days)
Population: Subjects in the ITT-LOCF patient population.
Measure: Count of Participants; unit: Participants
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%. 1.2 mg/ml | Placebo
Number analyzed (Participants) | 41 | 41 | 41
Participants | 18 | 17 | 12

4. Other Pre Specified Outcome: Mean Change in Schirmer's Test Score From Baseline to 84 Days (Visit 6) - Fellow Eye
Description: as for outcome 1
Time Frame: Visit 1 (baseline) to Visit 6 (84 Days)
Population: Subjects in the ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%. 1.2 mg/ml | Placebo
Number analyzed (Participants) | 41 | 41 | 41
mm | 7.9 (1.19) | 8.7 (1.18) | 4.8 (1.18)

5. Other Pre Specified Outcome: Mean Change in Schirmer's Test Score From Baseline to 28 Days (Visit 4) - Study Eye
Description: The Schirmer's test measures the amount of tears produced by numbing the eye and placing a paper strip in the eye for 5 minutes and distance of wetting was recorded following treatment of OC-01 or placebo. Schirmer's test scores range from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: Visit 1 (baseline) to Visit 4 (28 days)]
Population: Subjects in the ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%. 1.2 mg/ml | Placebo
Number analyzed (Participants) | 41 | 41 | 41
mm | 10.2 (1.42) | 11.4 (1.42) | 6.9 (1.42)

6. Other Pre Specified Outcome: Mean Change in Schirmer's Test Score From Baseline to 28 Days (Visit 4) - Fellow Eye
Description: as for outcome 1
Time Frame: Visit 1 (baseline) to Visit 4 (28 Days)
Population: Subjects in the ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%. 1.2 mg/ml | Placebo
Number analyzed (Participants) | 41 | 41 | 41
mm | 5.4 (1.36) | 9.2 (1.35) | 6.7 (1.35)

7. Other Pre Specified Outcome: Mean Change in Total Corneal Fluorescein Staining
Description: A standardized grading system of 0-3 is used for each of the five areas of the cornea (inferior, superior, nasal, temporal, central). Grade 0 will be specified when no staining is present. The total score ranges from 0-15. Lower scores indicate improvement.
Time Frame: Visit 1 (baseline) and Visit 5 (56 days)
Population: Subjects in the ITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%, 1.2 mg/ml | Placebo
Number analyzed (Participants) | 35 | 30 | 31
units on a scale | -3.3 (0.56) | -3.7 (0.6) | -3.2 (0.59)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug administration until the final study visit at Visit 6 (84 days).
Arm/Group | OC-01 0.1%, 0.6 mg/ml | OC-01 0.2%, 1.2 mg/ml | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 4/41 | 5/41 | 4/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC-01 0.1%, 0.6 mg/ml (N=41) | OC-01 0.2%, 1.2 mg/ml (N=41) | Placebo (N=41)
Ocular TEAEs (Eye disorders) | 4 (4) | 5 (5) | 4 (4) — Ocular TEAEs
Visual acuity reduced (Eye disorders) | 4 (4) | 3 (3) | 3 (3)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT03873246/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT03873246/SAP_001.pdf